CLINICAL TRIAL: NCT00638092
Title: A Randomised Controlled Trial of Iodide Supplementation in Preterm Infants With Follow-up at 2 Years
Brief Title: A Randomised Controlled Trial of Iodide Supplementation in Preterm Infants Follow-up at 2 Years
Acronym: I2S2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Dundee (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08/S0501/31; 2008-001024-31 (EudraCT Number); 08/S0501/31 (Other: REC Reference); 09/800/03 (Other Grant/Funding Number: NIHR EME)
Record Dates: First submitted 2008-03-14; First posted 2008-03-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Transient Hypothyroxinemia
Keywords: hypothyroxinemia; preterm infants; iodine; neurodevelopmental outcome; Iodine supplementation; Randomised controlled trial
MeSH Terms: interventions — Sodium Iodide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodine (Experimental): This is the hypothetical active arm
  Interventions: Drug: sodium iodide
- Placebo (Placebo Comparator): this is the hypothetical placebo
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: sodium iodide — sodium iodide 30 micrograms/kg/day, daily dose, from randomisation (within 42 hours of birth) to 34 corrected weeks gestation
  Arms: Iodine
Drug: Sodium Chloride — Sodium Chloride 30 micrograms/kg/day, daily dose, from randomisation (from within 42 hours of birth)to 34 corrected weeks gestation
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine whether iodide supplementation of neonates born under 31 weeks gestation improves neurodevelopment measured at two years of age.

DETAILED DESCRIPTION:
Iodine is essential for the synthesis of thyroxine, and thyroxine is essential for normal brain development in utero and for the first 2-3 years of life. The recommended iodine intake in parenteral nutrition regimens is 1 μg/kg/day and commercially available parenteral solutions for infants reflect these recommendations. In the absence of other iodine sources, infants are vulnerable to negative iodine balance and insufficiency. As many preterm infants are fed parenterally for prolonged periods with solutions which have been shown to be iodine-deficient, the I2S2 Trial was designed as a UK multicentre randomised controlled trial to establish whether iodine supplementation of preterm infants benefits neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* All infants born under 31 weeks gestation

Exclusion Criteria:

* Mother exposed to excess iodine during pregnancy or delivery

Ages: 1 Hour to 42 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1275 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Appreciable neurodevelopmental impairment at 2 years corrected age. As measured by the three main domains of the Bayley III score: i.e. cognitive score, language composite score and motor composite score. | at 2 years corrected age
  P ≤0.05 will be the level used to indicate statistical significance.Deaths and those infants with severe neurodevelopment disability will be scored 55 in the cognitive domain, 46 in the motor domain and 47 in the language domain. The primary outcome will be ordered as cognitive score, motor composite score and language composite score in all results presented.

SECONDARY OUTCOMES:
Blood levels of T4, TSH and TBG on day 7, 14, 28 and 34 weeks corrected age. | 2 years corrected age
Neurodevelopment impairment as a composite of death or a Bayley III score of <85 in any of the score's three main subsets domains: cognitive, language and motor composites. | 2 years corrected age
Neurodevelopmental impairment assessed as a difference between the iodine supplemented and placebo groups in each of the four subset scores of the Bayley III i.e. receptive communication, expressive communication, fine motor or gross motor. | 2 years corrected age
Type and severity of illness: necrotising enterocolitis | 2 years corrected age
  Type and severity of illness: necrotising enterocolitis
Type and severity of illness:persistent ductus arteriosus | 2 years corrected age
  Type and severity of illness:persistent ductus arteriosus
Type and severity of illness: respiratory distress | 2 years corrected age
  Type and severity of illness: respiratory distress
Type and severity of illness:chronic lung disease (need for oxygen at 36 weeks corrected age) | 2 years corrected age
  Type and severity of illness: chronic lung disease (need for oxygen at 36 weeks corrected age)
Cranial ultrasound changes | 2 years corrected age
  cranial ultrasound changes
Acquired infection | 2 years corrected age
  Acquired infection as indicated by medical notes during neonatal period
Cranial ultrasound changes | 2 years corrected age
  Type and severity of illness: necrotising enterocolitis, persistent ductus arteriosus, respiratory distress , chronic lung disease (need for oxygen at 36 weeks corrected age), cranial ultrasound changes, acquired infection; hearing and vision impairment; postnatal drug use (e.g. diamorphine, dexamethasone, dopamine, caffeine and indomethacin); nutritional status; BAPM level of care; highest recorded bilirubin levels; and death - immediate and underlying causes.
Hearing and vision impairment | 2 years corrected age
  Hearing and vision impairment as indicated by parental questionnaire
Postnatal drug use | 2 years corrected age
  diamorphine, dexamethasone, dopamine, caffeine and indomethacin
Nutritional status | 2 years corrected age
  Nutritional status collected on postnatal day 7, 14, 28 and 34 corrected weeks (as indicated by neonatal drug chart
BAPM level of care | 2 years corrected age
  BAPM level of care
Highest recorded bilirubin levels | 2 years corrected age
  highest recorded bilirubin levels; and death - immediate and underlying causes.
Death - immediate and underlying causes. | 2 years corrected age
  Death - immediate and underlying causes.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Williams, Dr, Study Director — University of Dundee; Peter Brocklehurst, Professor, Study Chair — UCL
Locations (19):
- United Kingdom (19):
  - Ninewells Hospital and Medical School, Dundee, Tayside
  - Royal Maternity Hospital, Belfast
  - Heartlands Hospital, Birmingham
  - University Hospital Coventry, Coventry
  - Derbyshire Childrens Hospital, Derby
  - Princess Royal Maternity Hospital, Glasgow
  - Southern General Hospital, Glasgow
  - Crosshouse Hospital, Kilmarnock
  - Leicester Royal Infirmary, Leicester
  - Altnagelvin Area Hospital, Londonderry
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Queen's Medical Centre, Nottingham
  - Royal Berkshire Hospital, Reading
  - Jessops Wing Hospital, Sheffield
  - University Hospital of North Tees, Stockton-on-Tees
  - Sunderland City Hospitals, Sunderland
  - Wishaw General Hospital, Wishaw

REFERENCES:
- [Background] Williams F, Hume R, Ogston S, Brocklehurst P, Morgan K, Juszczak E; I2S2 team. A summary of the iodine supplementation study protocol (I2S2): a UK multicentre randomised controlled trial in preterm infants. Neonatology. 2014;105(4):282-9. doi: 10.1159/000358247. Epub 2014 Feb 27. PMID 24576827
- See also: Supports programme of work — http://www.euthyroid.org